CLINICAL TRIAL: NCT01108445
Title: A Randomized Phase II Study of Afinitor (RAD001) vs. Sutent (Sunitinib) in Patients With Metastatic Non-Clear Cell Renal Cell Carcinoma (ASPEN)
Brief Title: Phase II Study of Afinitor vs. Sutent in Patients With Metastatic Non-Clear Cell Renal Cell Carcinoma
Acronym: ASPEN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Novartis (Industry); Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00020714; CRAD001L2402T (Other: Novartis)
Record Dates: First submitted 2010-04-20; First posted 2010-04-22 (Estimated); Results first posted 2016-06-20 (Estimated); Last update posted 2018-01-16 (Actual); Status verified 2017-09

CONDITIONS: Advanced Non-clear Cell Renal Cell Carcinoma
Keywords: cancer; kidney cancer; sutent; everolimus; renal cancer; papillary renal cell; chromophobe renal cell; papillary; chromophobe
MeSH Terms: conditions — Neoplasms; Kidney Neoplasms | interventions — Everolimus; Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- RAD001 (Active Comparator): Subjects in this treatment arm will receive everolimus/RAD001 10 mg orally once daily by mouth on days 1 through 42 for each 42 day cycle.
  Interventions: Drug: Everolimus
- Sunitinib (Active Comparator): Subjects in this treatment arm will take sunitinib 50 mg daily by mouth on days 1 through 28 of each 42 day cycle.
  Interventions: Drug: Sunitinib

INTERVENTIONS:
Drug: Everolimus — Subjects in this treatment arm will receive everolimusRAD001 10 mg orally once daily by mouth on days 1 through 42 for each 42 day cycle.
  Other Names: Afinitor, everolimus, RAD001
  Arms: RAD001
Drug: Sunitinib — 50 mg daily by mouth on days 1 through 28 of each 42 day cycle.
  Other Names: Sutent
  Arms: Sunitinib

SUMMARY:
To compare the anti-tumor activity of everolimus and sunitinib in subjects with metastatic renal cell carcinoma (mRCC) with non-clear cell pathology.

DETAILED DESCRIPTION:
This will be an international (USA, Canada, and UK) open-label, outpatient, multicenter, randomized study of treatment with RAD001 (everolimus (Afinitor®) or sunitinib (Sutent®) in subjects with mRCC and non-clear cell histology. Special emphasis is placed on papillary and chromophobe histologies while sarcomatoid clear cell variants, medullary, and collecting duct carcinomas will be excluded (see eligibility). Subjects may continue receiving study drugs until disease progression, unacceptable toxicities, or withdrawal of consent, for a maximum of 24 months. Continuation of study assigned treatment will be allowed beyond 24 months at the discretion of the sponsor. Stratification variables will include histology (papillary vs. chromophobe) and Motzer risk criteria (0, 1-2, and 3). Tumor progression will be assessed locally and by independent review, in strict accordance with Response Evaluation Criteria in Solid Tumors (RECIST 1.1) criteria measured every 12 weeks. At the time of progression, subjects will be taken off study other than simple administrative mortality follow-up. Primary pathologic samples and plasma/urine angiokine levels at baseline and over time will be collected and stored centrally for biomarker analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed advanced Renal Cell Carcinoma (RCC), with non-clear cell pathology.
2. RCC tumor tissue available for correlative sciences, from either primary or metastatic site or both.
3. At the time of screening, at least 4 weeks since prior palliative radiation therapy and/or major surgery, and resolution of all toxic effects of prior therapy to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE; version 4.0) Grade 1.
4. Subject must have radiographic evidence of metastatic disease with at least 1 measurable per RECIST 1.1 criteria (Attachment 1)].
5. Age > 18 years.
6. Adequate laboratory values
7. Karnofsky Performance Status ≥ 60 (Attachment 2).
8. Life expectancy of at least 3 months.
9. Written, signed, dated, and witnessed Institutional Review Board (IRB) or Institutional Ethics Committee (IEC) approved informed consent form (ICF) before any screening procedures are performed.

Exclusion Criteria:

1. Subjects with a history of or active central nervous system (CNS) metastases.
2. Prior systemic therapy for RCC, including mTOR and anti-angiogenic therapy, chemotherapy, biologic or experimental therapy.
3. Subjects with collecting duct, medullary, small cell, oncocytoma, or lymphoma-type pathology.
4. Subjects receiving known strong CYP3A4 isoenzyme inhibitors and/or inducers.
5. Major surgery, open biopsy, traumatic injury, or radiotherapy within 4 weeks of the screening visit.
6. Subjects who have not recovered from prior biopsy, surgery, traumatic injury, and/or radiation therapy.
7. Presence of a non-healing wound or ulcer.
8. Grade 3 hemorrhage within the past month.
9. Hypertension with systolic blood pressure of >180 mm Hg and/or diastolic pressure >100 mm Hg.
10. Subjects with American Heart Association (AHA) Class 2-4 heart disease or any history of congestive heart failure with an ejection fraction <50%, or history of unstable angina, myocardial infarction, coronary artery bypass graft, cerebrovascular accident, transient ischemic attack, or pulmonary embolism within 6 months of entry.
11. Diabetes mellitus with glycosylated hemoglobin A1c (HbgA1c) > 10% despite therapy.
12. A history of interstitial pneumonitis.
13. Subjects with active autoimmune disorder(s) being treated with immunosuppressive agents within 4 weeks prior to the screening visit.
14. Subjects receiving immunosuppressive agents and those with chronic viral/bacterial/fungal illnesses such as human immunodeficiency virus (HIV).
15. Patients who have receive immunization with attenuated live vaccines within one week of study entry or during study period.
16. Patients with active infection(s), active antimicrobial therapy or serious intercurrent illness.
17. History of other prior malignancy in past 5 years.
18. Pregnant or nursing women.
19. Major medical/psychiatric illness that, in the investigator's judgment, will substantially increase the risk associated with the subject's participation in this study, including inability to absorb oral medications and history of noncompliance to medical regimens.
20. Known hypersensitivity to any of the components in everolimus or sunitinib product
21. Subjects taking agents that significantly prolong the QTc interval are not eligible.
22. Proteinuria with a spot urine protein/creatinine ratio >2 or 24 hour urine protein >2 grams per 24 hours.
23. Severely impaired lung function as defined as spirometry and Carbon Monoxide Diffusing Capacity (DLCO) that is 50% of the normal predicted value and/or O2 saturation that is 88% or less at rest on room air.
24. Advanced liver disease such as cirrhosis or severe hepatic impairment (Child-Pugh class C).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2010-09; Primary Completion 2015-02 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Armstrong, MD, ScM, Principal Investigator — Duke University
Locations (18):
- United States (9):
  - University of Chicago, Chicago, Illinois
  - Indiana University Melvin and Bran Simon Cancer Center, Indianapolis, Indiana
  - Karmanos Cancer Institute/Wayne State University, Detroit, Michigan
  - Washington Univ in St. Louis-School of Medicine, St Louis, Missouri
  - Duke Univeristy Medical Center, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - SCRI, Nashville, Tennessee
  - The Vanderbilt Clinic, Henry-Joyce Cancer Center, Nashville, Tennessee
- Canada (3):
  - BC Cancer Agency, Vancouver, British Columbia
  - CancerCare Manitoba, Med Onc, Dept Hem and Onc, Winnipeg, Manitoba
  - London Health Sciences Center, London, Ontario
- United Kingdom (6):
  - Cambridge Cancer Trials Centre, Cambridge, England
  - The Royal Marsden NHS, London, England
  - The Christie Hospital NHS, Manchester, England
  - Weston Park Hospital, Sheffield, England
  - Churchill Hospital, Headington, Oxford
  - Beatson West Scotland Cancer Centre, Glasgow, Scottland

REFERENCES:
- [Derived] Aldin A, Besiroglu B, Adams A, Monsef I, Piechotta V, Tomlinson E, Hornbach C, Dressen N, Goldkuhle M, Maisch P, Dahm P, Heidenreich A, Skoetz N. First-line therapy for adults with advanced renal cell carcinoma: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 May 4;5(5):CD013798. doi: 10.1002/14651858.CD013798.pub2. PMID 37146227
- [Derived] Armstrong AJ, Halabi S, Eisen T, Broderick S, Stadler WM, Jones RJ, Garcia JA, Vaishampayan UN, Picus J, Hawkins RE, Hainsworth JD, Kollmannsberger CK, Logan TF, Puzanov I, Pickering LM, Ryan CW, Protheroe A, Lusk CM, Oberg S, George DJ. Everolimus versus sunitinib for patients with metastatic non-clear cell renal cell carcinoma (ASPEN): a multicentre, open-label, randomised phase 2 trial. Lancet Oncol. 2016 Mar;17(3):378-388. doi: 10.1016/S1470-2045(15)00515-X. Epub 2016 Jan 13. PMID 26794930
- [Derived] Winquist E, Rodrigues G. Open clinical uro-oncology trials in Canada. Can J Urol. 2012 Dec;19(6):6587-91. No abstract available. PMID 23228299

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 131 participants signed consent. 22 were screen failures. 1 withdrew consent prior to being randomized. 108 participant were randomized.
Period: Overall Study
Arm/Group | RAD001 | Sunitinib
Started | 57 | 51
Completed | 1 | 2
Not Completed | 56 | 49

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RAD001 | Sunitinib | Total
Number analyzed (Participants) | 57 | 51 | 108
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.9 (11.85) | 60.9 (15.3) | 61.4 (13.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 14 | 27
  Male | 44 | 37 | 81

OUTCOME MEASURES:

1. Primary Outcome: Anti-tumor Activity as Measured by Median Progression Free Survival Time
Description: The primary objective will be to compare the anti-tumor activity of everolimus and sunitinib in subjects with mRCC with non-clear cell pathology, as measured by progression-free survival (PFS) following treatment initiation according to RECIST 1.1 criteria. Progressive disease is defined as at least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression).
Time Frame: 24 Months
Measure: Median (80% Confidence Interval); unit: Months
Arm/Group | RAD001 | Sunitinib
Number analyzed (Participants) | 57 | 51
Months | 5.6 [5.5 to 6.0] | 8.3 [5.8 to 11.4]
Statistical Analysis 1: Comparison: RAD001 vs Sunitinib; Test type: Superiority or Other; p = 0.157, Log Rank; Hazard Ratio (HR) = 1.406

2. Secondary Outcome: Progression Free Survival Rates
Description: 6-, 12-, and 24-month rates of PFS in each arm will be compared for each treatment arm. Progressive disease is defined as at least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression).
Time Frame: 6, 12 and 24 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | RAD001 | Sunitinib
Number analyzed (Participants) | 57 | 51
percentage of participants
  6 Months | 40.3 [27.3 to 52.8] | 55.0 [40.1 to 67.7]
  12 Months | 17.0 [8.4 to 28.3] | 37.7 [24.1 to 51.2]
  24 Months | 9.3 [3.0 to 20.2] | 22.8 [11.7 to 36.1]

3. Secondary Outcome: PFS Expressed in Months
Description: Progression-free survival (PFS) expressed in months as compared to an historic control (interferon-treated clear cell RCC control arm from the sunitinib phase III study). Progressive disease is defined as at least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression).
Time Frame: 24 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | RAD001 | Sunitinib
Number analyzed (Participants) | 57 | 51
Months | 5.6 [4.4 to 6.1] | 8.3 [5.6 to 13.0]
Statistical Analysis 1: Comparison: RAD001; A comparison of the median PFS for RAD001 arm was compared to the 95% confidence interval(CI) of the median PFS of the historical control (HC). The null hypothesis was that there is no difference in the median PFS between the treatment arms and the historical control. If the median PFS is outside the 95%CI for the HC,it is determined there is statistical evidence that median PFS is different from the HC; Test type: Superiority or Other; Median PFS = 5.6 — The 95% CI for the HC was (4,6). If the median PFS for RAD001 is within the 95% CI for the HC, it is determined that there is not enough statistical evidence to say that the median PFS is different than the HC
Statistical Analysis 2: Comparison: Sunitinib; A comparison of the median PFS for Sunitinib arm was compared to the 95% confidence interval(CI) of the median PFS of the historical control (HC). The null hypothesis was that there is no difference in the median PFS between the treatment arms and the historical control. If the median PFS is outside the 95%CI for the HC,it is determined there is statistical evidence that median PFS is different from the HC; Test type: Superiority or Other; Median PFS = 8.3 — 95% CI for HC was(4,6). If the median PFS for Sunitinib is within the 95% CI for the HC,it is determined that there is not enough statistical evidence to say that the median PFS is different than the HC

4. Secondary Outcome: Overall Response Rate
Description: Defined as complete response [CR] and partial response [PR] by RECIST 1.1 criteria in each treatment arm.Overall Response Rate (ORR) = CR + PR. Complete Response (CR) is disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Partial Response (PR) is at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: 24 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | RAD001 | Sunitinib
Number analyzed (Participants) | 57 | 51
percentage of participants | 8.8 [1.4 to 16.1] | 17.6 [7.2 to 28.1]

5. Secondary Outcome: Percentage of Participants With Stable Disease (SD)
Description: Percentage of participants with stable disease during treatment is defined as stable disease [SD] by RECIST 1.1 criteria as calculated in each treatment arm. Stable Disease (SD) is defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Time Frame: Baseline to 36 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | RAD001 | Sunitinib
Number analyzed (Participants) | 57 | 51
percentage of participants | 59.6 [46.9 to 72.4] | 64.7 [51.6 to 77.8]
Statistical Analysis 1: Comparison: RAD001 vs Sunitinib; Test type: Superiority or Other; p = 0.589, Chi-squared

6. Secondary Outcome: 12 Week Clinical Benefit Rate as Percentage
Description: Rate of complete or partial response or stable disease by the RECIST 1.1 criteria lasting ≥ 12 weeks prior to progression. Benefit rate is defined as complete response [CR] and partial response [PR] and stable disease [SD] by RECIST 1.1 criteria in each treatment arm. Benefit rate = CR + PR + SD. Complete Response (CR) is disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Partial Response (PR) is at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Time Frame: Baseline to 36 months
Measure: Number (95% Confidence Interval); unit: percentage of particpants
Arm/Group | RAD001 | Sunitinib
Number analyzed (Participants) | 57 | 51
percentage of particpants | 24.6 [13.4 to 35.7] | 41.2 [27.7 to 54.7]
Statistical Analysis 1: Comparison: RAD001 vs Sunitinib; Test type: Superiority or Other; p = 0.066, Chi-squared

7. Secondary Outcome: Overall Survival Rates
Description: To compare overall survival (OS) rates at 6, 12, 24, and 36 months and over time in each treatment arm.
Time Frame: 6, 12, 24, 36 months
Measure: Number (95% Confidence Interval); unit: percentage probability
Arm/Group | RAD001 | Sunitinib
Number analyzed (Participants) | 57 | 51
percentage probability
  6 months | 83.5 [70.7 to 91.1] | 85.4 [71.8 to 92.8]
  12 months | 57.7 [43.0 to 69.8] | 74.7 [59.7 to 84.8]
  24 months | 40.8 [26.4 to 54.6] | 51.3 [35.1 to 65.3]
  36 months | 35.7 [20.6 to 51.0] | 46.2 [29.0 to 61.7]

8. Secondary Outcome: Best Tumor Shrinkage as a Percentile in Each Arm
Description: To compare the best tumor shrinkage as a percentile in each treatment arm. The percentile change at each follow up visit is calculated by measuring the percentage change in the Sum of lesion measurement from baseline. The best tumor shrinkage is lowest percentile change. A decrease is indicated by a negative percentage.
Time Frame: 24 months
Measure: Median (Inter-Quartile Range); unit: percentile decrease
Arm/Group | RAD001 | Sunitinib
Number analyzed (Participants) | 57 | 51
percentile decrease | -2.1 [-14.5 to 5.8] | -10.7 [-24.1 to 7.1]

9. Secondary Outcome: Median Duration of Response (CR, PR, and SD)
Description: To compare the median duration of response (CR, PR, and SD) in each treatment arm. According to RECIST 1.1, Complete Response (CR) is disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Partial Response (PR) is at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Time Frame: 24 months
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | RAD001 | Sunitinib
Number analyzed (Participants) | 57 | 51
months | 3.9 [2.8 to 9.1] | 8.3 [3.1 to 17.2]

10. Secondary Outcome: Median OS
Description: To compare the median OS in each treatment arm.
Time Frame: Up to 40 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | RAD001 | Sunitinib
Number analyzed (Participants) | 57 | 51
months | 13.2 [9.7 to 37.9] | 31.5 [14.8 to NA] — The upper limit of the 95% confidence interval was not calculable because an insufficient number of participants reached the event at the final time point for assessment.

11. Secondary Outcome: Time-to-new Metastatic Disease in Each Treatment Arm
Description: To compare the time-to-new metastatic disease in each treatment arm, defined from the date of first study agent administration to the onset of a new evaluable site of disease, excluding the primary site and all sites documented at baseline
Time Frame: 36 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | RAD001 | Sunitinib
Number analyzed (Participants) | 57 | 51
months | 19.4 [8.2 to 36] | 36 [11.4 to 36]

12. Secondary Outcome: Percentage of Participants With Adverse Events
Description: To assess toxicities associated with everolimus or sunitinib using NCI CTC version 4.0 criteria
Time Frame: 24 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | RAD001 | Sunitinib
Number analyzed (Participants) | 57 | 51
percentage of participants | 63.2 [50.6 to 75.7] | 80.4 [69.5 to 91.3]

13. Secondary Outcome: Change in Quality-of-life
Description: To compare change in quality-of-life, as measured by the FACT-KSI scale at baseline and cycle 3 day 1 per subject in each treatment arm. Functional Assessment of Cancer Therapy Kidney Symptom Index. FKSI is a questionnaire for FACT-Kidney Symptom Index used to assess QoL/participant-reported outcomes for participants diagnosed with renal cell cancer. The FKSI contained 15 questions each ranging from 0 (not at all) to 4 (very much) so that FKSI ranged between 0-60 where higher scores reflects better functioning and fewer symptoms.
Time Frame: baseline, cycle 3 day 1
Population: All participants who completed the cycle 3 day 1 visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | RAD001 | Sunitinib
Number analyzed (Participants) | 30 | 31
units on a scale | -3.5 (9.61) | -0.9 (7.19)

14. Secondary Outcome: Change in Quality-of-life
Description: To compare change in quality-of-life, as measured by the FACT-KSI scale at baseline and cycle 6 day1 per subject in each treatment arm. Functional Assessment of Cancer Therapy Kidney Symptom Index. FKSI is a questionnaire for FACT-Kidney Symptom Index used to assess QoL/participant-reported outcomes for participants diagnosed with renal cell cancer. The FKSI contained 15 questions each ranging from 0 (not at all) to 4 (very much) so that FKSI ranged between 0-60 where higher scores reflects better functioning and fewer symptoms.
Time Frame: baseline, cycle 6 day 1
Population: All participants who completed the cycle 6 day 1 visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | RAD001 | Sunitinib
Number analyzed (Participants) | 13 | 17
units on a scale | -4.4 (6.37) | -2.1 (6.69)

15. Secondary Outcome: Change in Quality-of-life
Description: To compare change in quality-of-life, as measured by the FACT-KSI scale at baseline and end of treatment per subject in each treatment arm. Functional Assessment of Cancer Therapy Kidney Symptom Index. FKSI is a questionnaire for FACT-Kidney Symptom Index used to assess QoL/participant-reported outcomes for participants diagnosed with renal cell cancer. The FKSI contained 15 questions each ranging from 0 (not at all) to 4 (very much) so that FKSI ranged between 0-60 where higher scores reflects better functioning and fewer symptoms.
Time Frame: baseline, up to 40 months
Population: All participants who completed the End of treatment visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | RAD001 | Sunitinib
Number analyzed (Participants) | 32 | 30
units on a scale | -6.6 (7.83) | -6.4 (10.04)

16. Other Pre Specified Outcome: Clinical Measures of Response and PFS With Baseline and Time-dependent Levels of Biomarkers
Description: To correlate clinical measures of response and PFS with baseline and time-dependent levels of biomarkers. These biomarkers include plasma angiokine levels, tissue immunohistochemical and genomic profiles, copy number as assessed by array-based comparative genomic hybridization (CGH), and known mutations in non-clear cell RCC
Time Frame: 36 months
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Changes in Copy Number, RNA Expression, and Immunohistochemical Profiles
Description: To evaluate in an exploratory fashion changes in copy number, RNA expression, and immunohistochemical profiles by microarray between primary non-clear cell RCC tumors and metastatic samples
Time Frame: 36 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Baseline to 40 months
Arm/Group | RAD001 | Sunitinib
Serious Adverse Events (participants affected / at risk) | 36/57 | 41/51
Other Adverse Events (participants affected / at risk) | 57/57 | 51/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RAD001 (N=57) | Sunitinib (N=51)
Abdominal pain (Gastrointestinal disorders) | 2 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 2 | 2
Diarrhoea (Gastrointestinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 1 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 1 | 3
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Disease progression (General disorders) | 2 | 1
Mucosal inflammation (General disorders) | 1 | 0
Multi-organ failure (General disorders) | 1 | 0
Pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 1
Anal abscess (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Haemoglobin decreased (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 1 | 0
Haemorrhagic stroke (Nervous system disorders) | 1 | 0
Spinal cord compression (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 1
Delirium (Psychiatric disorders) | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 1
Nephropathy toxic (Renal and urinary disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 2 | 2
Renal impairment (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 5 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1
Embolism arterial (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 2
Embolism venous (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RAD001 (N=57) | Sunitinib (N=51)
Anaemia (Blood and lymphatic system disorders) | 16 | 14
Leukopenia (Blood and lymphatic system disorders) | 2 | 4
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 5
Thrombocytopenia (Blood and lymphatic system disorders) | 7 | 12
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 0 | 1
Palpitations (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 1
Cardiac flutter (Cardiac disorders) | 0 | 1
Left ventricular hypertrophy (Cardiac disorders) | 0 | 1
Ear disorder (Ear and labyrinth disorders) | 1 | 0
Ear pain (Ear and labyrinth disorders) | 2 | 0
Ear pruritus (Ear and labyrinth disorders) | 1 | 0
Otorrhoea (Ear and labyrinth disorders) | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 1
Hyperthyroidism (Endocrine disorders) | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 3
Cataract (Eye disorders) | 1 | 0
Conjunctivitis (Eye disorders) | 1 | 0
Dry eye (Eye disorders) | 2 | 2
Eye discharge (Eye disorders) | 1 | 0
Eye irritation (Eye disorders) | 1 | 0
Eye pain (Eye disorders) | 1 | 0
Periorbital oedema (Eye disorders) | 2 | 2
Vision blurred (Eye disorders) | 2 | 0
Conjunctival hyperaemia (Eye disorders) | 0 | 1
Conjunctival oedema (Eye disorders) | 0 | 1
Conjunctival pallor (Eye disorders) | 0 | 1
Eye swelling (Eye disorders) | 0 | 1
Eyelid oedema (Eye disorders) | 0 | 1
Glaucoma (Eye disorders) | 0 | 1
Lacrimation increased (Eye disorders) | 0 | 3
Photopsia (Eye disorders) | 0 | 1
Vitreous floaters (Eye disorders) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 2 | 3
Abdominal pain (Gastrointestinal disorders) | 7 | 7
Abdominal pain lower (Gastrointestinal disorders) | 1 | 2
Abdominal pain upper (Gastrointestinal disorders) | 3 | 5
Ascites (Gastrointestinal disorders) | 1 | 1
Cheilitis (Gastrointestinal disorders) | 4 | 0
Constipation (Gastrointestinal disorders) | 10 | 15
Diarrhoea (Gastrointestinal disorders) | 15 | 34
Dry mouth (Gastrointestinal disorders) | 4 | 5
Dyspepsia (Gastrointestinal disorders) | 5 | 11
Dysphagia (Gastrointestinal disorders) | 1 | 1
Faeces discoloured (Gastrointestinal disorders) | 1 | 1
Flatulence (Gastrointestinal disorders) | 1 | 6
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 8
Gingival pain (Gastrointestinal disorders) | 1 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 0
Lip swelling (Gastrointestinal disorders) | 1 | 0
Mouth ulceration (Gastrointestinal disorders) | 5 | 1
Nausea (Gastrointestinal disorders) | 26 | 36
Oral pain (Gastrointestinal disorders) | 2 | 4
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 27 | 14
Tongue blistering (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 13 | 17
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1
Anal inflammation (Gastrointestinal disorders) | 0 | 1
Dental caries (Gastrointestinal disorders) | 0 | 1
Gingival bleeding (Gastrointestinal disorders) | 0 | 1
Gingival hypertrophy (Gastrointestinal disorders) | 0 | 1
Glossodynia (Gastrointestinal disorders) | 0 | 2
Haematochezia (Gastrointestinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 2
Lip pain (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 3
Reflux oesophagitis (Gastrointestinal disorders) | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 1 | 2
Chest pain (General disorders) | 2 | 0
Chills (General disorders) | 4 | 3
Fatigue (General disorders) | 33 | 31
Hernia (General disorders) | 1 | 0
Influenza like illness (General disorders) | 3 | 2
Irritability (General disorders) | 1 | 1
Local swelling (General disorders) | 1 | 0
Mucosal inflammation (General disorders) | 13 | 12
Non-cardiac chest pain (General disorders) | 3 | 1
Oedema (General disorders) | 1 | 1
Oedema peripheral (General disorders) | 15 | 8
Pain (General disorders) | 4 | 5
Pyrexia (General disorders) | 8 | 4
Chest discomfort (General disorders) | 0 | 1
Early satiety (General disorders) | 0 | 1
Impaired healing (General disorders) | 0 | 1
Hepatotoxicity (Hepatobiliary disorders) | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1
Drug hypersensitivity (Immune system disorders) | 0 | 1
Seasonal allergy (Immune system disorders) | 0 | 1
Blister infected (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 1
Cystitis (Infections and infestations) | 1 | 0
Ear infection (Infections and infestations) | 4 | 1
Folliculitis (Infections and infestations) | 1 | 2
Furuncle (Infections and infestations) | 1 | 1
Hepatitis B (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 1
Localised infection (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 2 | 1
Lung infection (Infections and infestations) | 1 | 0
Lymph gland infection (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 3 | 0
Paronychia (Infections and infestations) | 2 | 1
Pneumonia (Infections and infestations) | 1 | 1
Rash pustular (Infections and infestations) | 1 | 1
Respiratory tract infection (Infections and infestations) | 1 | 1
Rhinitis (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 2 | 1
Soft tissue infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 4
Candidiasis (Infections and infestations) | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 1
Hand-foot-and-mouth disease (Infections and infestations) | 0 | 1
Oral candidiasis (Infections and infestations) | 0 | 1
Peritonsillar abscess (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 1
Skin infection (Infections and infestations) | 0 | 3
Tooth abscess (Infections and infestations) | 0 | 2
Tooth infection (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 2
Urosepsis (Infections and infestations) | 0 | 1
Viral infection (Infections and infestations) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 3
Procedural pain (Injury, poisoning and procedural complications) | 2 | 0
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0
Heart injury (Injury, poisoning and procedural complications) | 0 | 1
Joint sprain (Injury, poisoning and procedural complications) | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 1
Post procedural swelling (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 2 | 5
Aspartate aminotransferase increased (Investigations) | 7 | 10
Blood alkaline phosphatase increased (Investigations) | 3 | 3
Blood cholesterol increased (Investigations) | 7 | 1
Blood creatine increased (Investigations) | 2 | 0
Blood creatinine increased (Investigations) | 6 | 9
Blood glucose increased (Investigations) | 1 | 0
Blood magnesium decreased (Investigations) | 1 | 0
Blood phosphorus decreased (Investigations) | 1 | 0
Blood potassium decreased (Investigations) | 1 | 1
Blood triglycerides increased (Investigations) | 3 | 0
Blood urea increased (Investigations) | 1 | 3
Chest X-ray abnormal (Investigations) | 1 | 0
Glomerular filtration rate decreased (Investigations) | 1 | 4
Haemoglobin decreased (Investigations) | 1 | 1
Liver function test abnormal (Investigations) | 2 | 2
Low density lipoprotein increased (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 3 | 8
Weight decreased (Investigations) | 10 | 7
Weight increased (Investigations) | 1 | 1
Activated partial thromboplastin time prolonged (Investigations) | 0 | 1
Aspartate aminotransferase (Investigations) | 0 | 2
Bacterial test positive (Investigations) | 0 | 1
Blood albumin decreased (Investigations) | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 3
Blood calcium decreased (Investigations) | 0 | 1
Blood ketone body increased (Investigations) | 0 | 1
Blood lactate dehydrogenase increased (Investigations) | 0 | 3
Blood lactic acid increased (Investigations) | 0 | 1
Blood pressure increased (Investigations) | 0 | 4
Blood thyroid stimulating hormone increased (Investigations) | 0 | 1
Clostridium test positive (Investigations) | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 0 | 1
Haptoglobin decreased (Investigations) | 0 | 1
Lipase increased (Investigations) | 0 | 2
Lymphocyte count decreased (Investigations) | 0 | 1
Mean cell haemoglobin increased (Investigations) | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 8
Protein total decreased (Investigations) | 0 | 1
Protein total increased (Investigations) | 0 | 1
Transaminases increased (Investigations) | 0 | 1
Urine output decreased (Investigations) | 0 | 1
White blood cell count decreased (Investigations) | 0 | 8
Decreased appetite (Metabolism and nutrition disorders) | 15 | 30
Dehydration (Metabolism and nutrition disorders) | 2 | 4
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0
Gout (Metabolism and nutrition disorders) | 2 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 7 | 4
Hyperkalaemia (Metabolism and nutrition disorders) | 3 | 4
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 | 0
Hypermagnesaemia (Metabolism and nutrition disorders) | 1 | 2
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 8 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 3
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 5 | 7
Hypophosphataemia (Metabolism and nutrition disorders) | 3 | 5
Acidosis (Metabolism and nutrition disorders) | 0 | 1
Hyperammonaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperamylasaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperlipasaemia (Metabolism and nutrition disorders) | 0 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 1
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 12
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 15
Bone pain (Musculoskeletal and connective tissue disorders) | 3 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 5 | 7
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 2
Muscle mass (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 6 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 7
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Soft tissue disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle swelling (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 2
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ageusia (Nervous system disorders) | 1 | 1
Dizziness (Nervous system disorders) | 3 | 6
Dysgeusia (Nervous system disorders) | 18 | 25
Headache (Nervous system disorders) | 6 | 5
Lethargy (Nervous system disorders) | 9 | 10
Loss of consciousness (Nervous system disorders) | 1 | 0
Migraine (Nervous system disorders) | 1 | 1
Neuropathy peripheral (Nervous system disorders) | 3 | 3
Paraesthesia (Nervous system disorders) | 2 | 1
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0
Asterixis (Nervous system disorders) | 0 | 1
Disturbance in attention (Nervous system disorders) | 0 | 1
Dysarthria (Nervous system disorders) | 0 | 1
Encephalomalacia (Nervous system disorders) | 0 | 1
Hepatic encephalopathy (Nervous system disorders) | 0 | 1
Hyperaesthesia (Nervous system disorders) | 0 | 1
Neurotoxicity (Nervous system disorders) | 0 | 1
Parosmia (Nervous system disorders) | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Depressed mood (Psychiatric disorders) | 1 | 1
Depression (Psychiatric disorders) | 2 | 3
Insomnia (Psychiatric disorders) | 6 | 3
Mental status changes (Psychiatric disorders) | 1 | 1
Mood altered (Psychiatric disorders) | 1 | 1
Sleep disorder (Psychiatric disorders) | 2 | 1
Anxiety (Psychiatric disorders) | 0 | 8
Confusional state (Psychiatric disorders) | 0 | 1
Dysphoria (Psychiatric disorders) | 0 | 1
Emotional distress (Psychiatric disorders) | 0 | 1
Restlessness (Psychiatric disorders) | 0 | 1
Bladder hypertrophy (Renal and urinary disorders) | 1 | 0
Bladder spasm (Renal and urinary disorders) | 1 | 0
Cystitis noninfective (Renal and urinary disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 2 | 2
Haematuria (Renal and urinary disorders) | 3 | 5
Micturition urgency (Renal and urinary disorders) | 2 | 0
Nocturia (Renal and urinary disorders) | 2 | 0
Pollakiuria (Renal and urinary disorders) | 6 | 1
Proteinuria (Renal and urinary disorders) | 1 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 3
Urinary tract pain (Renal and urinary disorders) | 2 | 1
Azotaemia (Renal and urinary disorders) | 0 | 1
Chromaturia (Renal and urinary disorders) | 0 | 1
Renal impairment (Renal and urinary disorders) | 0 | 1
Renal tubular necrosis (Renal and urinary disorders) | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 1
Urine flow decreased (Renal and urinary disorders) | 0 | 1
Oedema genital (Reproductive system and breast disorders) | 1 | 0
Perineal pain (Reproductive system and breast disorders) | 1 | 0
Scrotal swelling (Reproductive system and breast disorders) | 1 | 0
Breast discomfort (Reproductive system and breast disorders) | 0 | 1
Genital rash (Reproductive system and breast disorders) | 0 | 2
Pruritus genital (Reproductive system and breast disorders) | 0 | 1
Scrotal oedema (Reproductive system and breast disorders) | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 25 | 8
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 21 | 9
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 11 | 7
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 | 1
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 5 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 4
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 4
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 11 | 7
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 3 | 4
Hair colour changes (Skin and subcutaneous tissue disorders) | 1 | 2
Hair growth abnormal (Skin and subcutaneous tissue disorders) | 1 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 1 | 0
Onychoclasis (Skin and subcutaneous tissue disorders) | 1 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 1 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 8 | 21
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 9 | 7
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 18 | 11
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 6 | 2
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0
Skin reaction (Skin and subcutaneous tissue disorders) | 1 | 2
Skin toxicity (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Cold sweat (Skin and subcutaneous tissue disorders) | 0 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 3
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 3
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 0 | 1
Plantar erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Purpura (Skin and subcutaneous tissue disorders) | 0 | 1
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 1
Scab (Skin and subcutaneous tissue disorders) | 0 | 1
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 1
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 2
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 1
Yellow skin (Skin and subcutaneous tissue disorders) | 0 | 3
Deep vein thrombosis (Vascular disorders) | 1 | 1
Flushing (Vascular disorders) | 3 | 1
Hot flush (Vascular disorders) | 2 | 3
Hypertension (Vascular disorders) | 6 | 23
Hypotension (Vascular disorders) | 1 | 4
Thrombophlebitis superficial (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less